CLINICAL TRIAL: NCT00165698
Title: Efficacy and Safety Study on Menatetrenone in the Treatment of Postmenopausal Osteoporosis Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Takao Ishii, Asia regulatory affaires, Eisai Co., Ltd.
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS-012 (GLA-CHN-05-01)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal; osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: menatetranone
- 2 (Active Comparator)
  Interventions: Drug: alfacalcidol

INTERVENTIONS:
Drug: menatetranone — 15 mg three times a day orally for 12 months
  Arms: 1
Drug: alfacalcidol — 0.25 μg twice a day orally for 12 months
  Arms: 2

SUMMARY:
To determine the effect and safety of menatetrenone on treatment of postmenopausal osteoporosis comparing with alfacalcidol.

ELIGIBILITY:
Inclusion criteria :

* Postmenopausal women with menopause duration more than 5 years and with age between 45-75 years old (menopausal age ≥40), or if hysterectomy operated before natural menopause, the age of women between 60-75 years old.
* Subject with BMD (L2-4 or neck of femur) being more than 2 Standard Deviation (SD) below the young female adult mean (According to the standard of each center)
* BMI between 18 kg/m2-30 kg/m2.
* The anatomic structure of lumbar spine must be available for Dual-energy X-ray Absorptiometry (DEXA) examination, patient with serious scoliosis, bone trauma or sequela after orthopedics surgery, which makes BMD measurement difficult, should be excluded
* Subject who have given informed consent prior to participation in the trial and who undertake to comply with the protocol.

Exclusion Criteria

* Subject with conditions that are considered to effect osteoporosis, such as clear definite diabetes mellitus, rheumatoid arthritis, rheumatoid arthritis, hyperparathyroidism or other bone metabolic diseases.
* Subjects who have received treatment with active-type vitamin D3 preparation, other vitamin D preparations (>1000IU per day）, calcitonin, corticosteroid hormone, androgen, estrogen, other hormone, vitamin K preparation, in the 3 months prior to inanition of this study; Subjects who have received treatment with bisphosphonate preparation or Sodium Fluoride in the 1 year prior to inanition of this study; Subjects who have received treatment with Selective Estrogen Receptor Modulator (SERM) in the 6 months prior to inanition of this study
* Concurrent serious renal disease, hepatic disease, uncontrolled hypertension （≥150/100mmHg）, symptomatic ischemic heart disease, cerebral infarction or arteriosclerosis obliterans.
* Cancer history within 5 years.
* Subjects who take antacid containing aluminum in the preparation, warfarin or thrombolytic agents.
* Subject with any known abnormality in laboratory tests, which is deemed to be clinically significant by the investigator, which include:
* Serum alkaline phosphatace (ALP) > upper normal limit 10% (calculated according to the range of normal values of each center);
* Glutamic Oxalacetic Transaminase (AST)/ Glutamic Pyruvic Transaminase (ALT) > upper normal limit 50％(calculated according to the range of normal values of each center);
* Serum creatinine >1.5mg/dL (133μmol/L);
* Blood-fasting sugar ≥ 7mmol/L (126mg/L)
* Inability of subject to return for scheduled visits or to comply with any other aspect of the protocol.
* Subject who, in the opinion of the investigator, are poor medical candidates or pose any other risk for therapy with an investigational drug.

Ages: 45 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Di, Study Director — Eisai China Inc.
Locations (5):
- China (5):
  - Beijing Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Hua Dong Hospital, Shanghai
  - The Sixth People's Hospital affiliated to Shanghai Jiaopong University, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Menatetrenone: 15 mg t.i.d. orally for 12 months
- Alfacalcidol: 0.25 μg b.i.d. orally for 12 months
Period: Overall Study
Arm/Group | Menatetrenone | Alfacalcidol
Started | 120 | 120
Completed | 112 | 105
Not Completed | 8 | 15
Not completed — Adverse Event | 2 | 10
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Not Taken/Lost the medicine | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menatetrenone | Alfacalcidol | Total
Number analyzed (Participants) | 112 | 108 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline Participants are Full Anaylsis Set (FAS) Population
  years | 64.6 (6.1) | 64.2 (6.3) | 64.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 108 | 220
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Race
  participants
    Asian | 112 | 108 | 220
Region of Enrollment [Number; unit: participants]
  China | 112 | 108 | 220

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density BMD (Percentage) Change in Lumber Spine After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Full Range); unit: percentage of BMD
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 105
percentage of BMD | 1.22 [-5.35 to 14.14] | 2.17 [-15.13 to 38.23]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.26, Symbols rank sum test

2. Primary Outcome: Bone Mineral Density BMD (Percentage) Change in Collum Femoris After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Full Range); unit: percentage of BMD
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 105
percentage of BMD | 0.76 [-18.51 to 19.46] | 0.00 [-15.84 to 13.80]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.19, Symbols rank sum test

3. Primary Outcome: Bone Mineral Density BMD (Percentage) Change in Trochiter After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Full Range); unit: percentage of BMD
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 105
percentage of BMD | 2.66 [-31.69 to 87.34] | 1.76 [-38.60 to 74.76]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.31, Symbols rank sum test

4. Secondary Outcome: Bone Mineral Content BMC (Percentage) Change in Lumber Spine After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Full Range); unit: percentage of BMC
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 103
percentage of BMC | 2.39 [-9.97 to 21.59] | 2.81 [-16.88 to 19.84]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.869, symbols rank sum test

5. Secondary Outcome: Bone Mineral Content BMC (Percentage) Change in Collum Femoris After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Full Range); unit: percentage of BMC
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 103
percentage of BMC | 1.58 [-12.50 to 29.63] | 0.95 [-21.24 to 15.71]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.174, symbols rank sum test

6. Secondary Outcome: Bone Biomarker Osteocalcin (OC) Percentage Change After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Inter-Quartile Range); unit: percentage of OC
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 104
percentage of OC | -38.67 [-67.26 to 1.33] | -25.77 [-65.66 to 57.48]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.000, symbols rank sum test

7. Secondary Outcome: Bone Biomarker Undercarboxylated Osteocalcin (UCOC) Percentage Change After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Inter-Quartile Range); unit: percentage of UCOC
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 104
percentage of UCOC | -82.27 [-97.27 to 676.60] | -34.83 [-92.07 to 950.00]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.000, symbols rank sum test

8. Secondary Outcome: Bone Biomarker Undercarboxylated Osteocalcin/Osteocalcin (UCOC/OC) Percentage Change After 12 Months
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Median (Inter-Quartile Range); unit: percentage of UCOC/OC
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 104
percentage of UCOC/OC | -70.64 [-94.49 to 1185.50] | -8.47 [-85.68 to 610.61]
Statistical Analysis 1: Comparison: Menatetrenone vs Alfacalcidol; Test type: Superiority or Other; p = 0.000, symbols rank sum test

9. Secondary Outcome: New Fracture and Fall
Time Frame: 12 months
Population: Per Protocol Set (PPS)
Measure: Number; unit: participants
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 105
participants
  fracture | 2 | 4
  fall | 13 | 10

10. Secondary Outcome: Height (Meter)
Time Frame: Baseline and 12 months
Population: Per Protocol Set (PPS)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Menatetrenone | Alfacalcidol
Number analyzed (Participants) | 108 | 105
meters
  Baseline | 1.54 (0.05) | 1.55 (0.05)
  At 12 months | 1.54 (0.06) | 1.55 (0.05)

ADVERSE EVENTS:
Description: Safety Population
Arm/Group | Menatetrenone | Alfacalcidol
Serious Adverse Events (participants affected / at risk) | 8/117 | 6/118
Other Adverse Events (participants affected / at risk) | 81/117 | 74/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menatetrenone (N=117) | Alfacalcidol (N=118)
Skin damage (Skin and subcutaneous tissue disorders) | 1 | 0
Bone fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Tendon damage (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Parathyroid malignant tumor (Endocrine disorders) | 0 | 1
NTT (Endocrine disorders) | 1 | 0
Goiter (Endocrine disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Chest distress (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Angina (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Breast cancer (Reproductive system and breast disorders) | 0 | 1
Nerve sheath tumor surgery (Surgical and medical procedures) | 0 | 1
Uterus resection (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menatetrenone (N=117) | Alfacalcidol (N=118)
Abnormal on skin and its subsidiary tissues (Skin and subcutaneous tissue disorders) | 7 | 5
Musculoskeletal system abnormalities (Musculoskeletal and connective tissue disorders) | 20 | 18
Central and peripheral nervous system abnormalities (Nervous system disorders) | 10 | 9
Gastrointestinal disorders (Gastrointestinal disorders) | 37 | 32
Abnormal liver system (Hepatobiliary disorders) | 7 | 6
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 8 | 3
Abnormal Cardiovascular system (Cardiac disorders) | 16 | 10
Heart rate and rhythm disorders (Cardiac disorders) | 9 | 8
Respiratory abnormalities (Respiratory, thoracic and mediastinal disorders) | 24 | 35
Urinary system abnormalities (Renal and urinary disorders) | 12 | 12
Systemic anomalies (General disorders) | 8 | 6
Others (General disorders) | 27 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No